CLINICAL TRIAL: NCT01583881
Title: Sympathetic Renal Denervation in Heart Failure With Normal LV Ejection Fraction: Denervation of the renAl sympathetIc nerveS in hearT Failure With nOrmal Lv Ejection Fraction
Brief Title: Denervation of the renAl sympathetIc nerveS in hearT Failure With nOrmal Lv Ejection Fraction
Acronym: DIASTOLE
Status: Terminated | Phase: Phase 2 / Phase 3 | Type: Interventional
Why Stopped: Slow inclusion
Sponsor: UMC Utrecht (Other)
Collaborators: VU University of Amsterdam (Other)
Responsible Party: Principal Investigator, Michiel Voskuil, MD, PhD, MD. PhD., UMC Utrecht
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 12-046
Record Dates: First submitted 2012-04-19; First posted 2012-04-24 (Estimated); Last update posted 2021-05-03 (Actual); Status verified 2021-04

CONDITIONS: Diastolic Heart Failure; Hypertension
Keywords: Patients with diastolic heart failure and hypertension
MeSH Terms: conditions — Heart Failure, Diastolic; Hypertension

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Renal denervation (Experimental): Renal denervation
  Interventions: Procedure: renal denervation
- control (No Intervention): No intervention

INTERVENTIONS:
Procedure: renal denervation — Renal denervation
  Arms: Renal denervation

SUMMARY:
Increasing evidence suggests an important role of activation of the sympathetic nervous system (SNS) in the clinical phenomena of heart failure with normal left ventricular ejection fraction and hypertension. The current study aims to evaluate efficacy and safety of renal sympathetic denervation for the modulation of the SNS in patients with heart failure with normal LV ejection fraction.

DETAILED DESCRIPTION:
Rationale: Increasing evidence suggests an important role of activation of the sympathetic nervous system (SNS) in the clinical phenomena of heart failure with normal left ventricular ejection fraction and hypertension. Moreover, sympathetic activation of the kidneys is directly proportional related to the severity of the heart failure state. Therapeutic renal denervation (PRDN), the deliberate disruption of the nerves connecting the kidneys with the central nervous system, has been shown to be an effective means of modulating elevated SNS activity. The current study aims to evaluate efficacy and safety of renal sympathetic denervation for the modulation of the SNS in patients with heart failure with normal LV ejection fraction.

Objective: Primary objectives: To investigate the efficacy of PRDN by means of pulsed wave Doppler echocardiographic parameters in patients diagnosed with HFNEF and hypertension. Secondary objectives: to investigate the safety of PRDN in patients with heart failure with normal LV ejection fraction and hypertension and to compare changes in the following parameters in patients with HFNEF and hypertension after PRDN: LV mass, LV volume, LA volume, LVEF, MIBG-uptake and -washout, BNP levels, blood pressure, heart rate variability, exercise capacity and quality of life.

Study design: Multicentre, prospective, randomised controlled trial. 60 patients will be randomly allocated in a one-to-one ratio to undergo renal denervation with previous treatment (n=30) or to maintain previous treatment alone (n=30) at 2 participating centres. Randomisation will be done with sealed envelopes.

Study population: Patients diagnosed with heart failure with normal LV ejection fraction and treated for hypertension. Patients should have a stable drug regimen, with at least 2 antihypertensive agents. This drug regimen should be expected to be maintained for at least 6 months.

￼￼￼￼￼￼￼￼￼Endpoints: The efficacy of PRDN will be evaluated primarily using echocardiographic parameters. Also, safety of PRDN on major and minor adverse events, LV mass, LV and LA dimensions, MIBG uptake and clinical endpoints will be evaluated.

ELIGIBILITY:
Inclusion Criteria:

* Individual is diagnosed with heart failure with a normal LV ejection fraction. The diagnosis of HFNEF requires the following conditions to be satisfied:

  * signs or symptoms of heart failure;
  * normal or mildly abnormal systolic LV function (LVEF ≥ 50%);
  * evidence of diastolic LV dysfunction.
* Individual should fulfill the diagnostic WHO criteria for hypertension: SBP > 140 mmHg and/or DBP > 90 mmHg, and is treated with at least 2 antihypertensive drugs. This treatment is expected to be maintained for at least 6 months. Using this regimen the blood pressure should be adequately controlled (< 140/90mmHg by 24 hour ambulatory BP measurement).
* Individual is adhering to a stable drug regimen HFNEF, with no changes for a minimum of 2 weeks prior to enrollment, and which is expected to be maintained for at least 6 months.
* Individual is ≥ 18 years of age.

Exclusion Criteria:

* Known secondary cause of hypertension
* Anatomy not eligible for renal denervation
* Systolic heart failure (LVEF < 50%)
* Individual has an estimated glomerular filtration rate (eGFR) of < 30mL/min/1.73m2, using the MDRD calculation.
* Individual has any serious medical condition, which in the opinion of the investigator, may adversely affect the safety and/or effectiveness of the participant or the study (i.e., patients with clinically significant peripheral vascular disease, abdominal aortic aneurysm, bleeding disorders such as thrombocytopenia, haemophilia, significant anaemia, or arrhythmias such as atrial fibrillation).
* Individual is pregnant, nursing or planning to be pregnant.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2012-04-01 (Actual); Primary Completion 2016-06-01 (Actual); Study Completion 2016-07-01 (Actual)

PRIMARY OUTCOMES:
Change from baseline E/E' at 12 months | 12 months after treatment
  Echocardiography will be used to measure the E/E'

SECONDARY OUTCOMES:
Number of participants with adverse events | 1 year

CONTACTS AND LOCATIONS:
Overall Officials: Michiel Voskuil, MD, PhD, Principal Investigator — UMC Utrecht
Locations (2):
- Netherlands (2):
  - VUmc, Amsterdam
  - UMC Utrecht, Utrecht

REFERENCES:
- [Derived] Verloop WL, Beeftink MM, Nap A, Bots ML, Velthuis BK, Appelman YE, Cramer MJ, Agema WR, Scholtens AM, Doevendans PA, Allaart CP, Voskuil M. Renal denervation in heart failure with normal left ventricular ejection fraction. Rationale and design of the DIASTOLE (DenervatIon of the renAl Sympathetic nerves in hearT failure with nOrmal Lv Ejection fraction) trial. Eur J Heart Fail. 2013 Dec;15(12):1429-37. doi: 10.1093/eurjhf/hft119. Epub 2013 Jul 24. PMID 23883653